CLINICAL TRIAL: NCT06710184
Title: Aspirin Versus Aspirin and Fondaparinux Prior to Early Invasive Strategy in Patients With NSTEMI
Brief Title: Treatment With Aspirin Alone Versus Aspirin in Combination With Fondaparinux Before Early Coronary Assessment in Patients With Non-ST-Elevation Myocardial Infarction
Acronym: FOXY
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danske Regioner (Other); Aalborg University Hospital (Other); Odense University Hospital (Other); Rigshospitalet, Denmark (Other); Randers Regional Hospital (Other); Viborg Regional Hospital (Other); Gødstrup Hospital (Other); Sydvestjysk Hospital Esbjerg (Unknown); Lillebaelt Hospital, Kolding and Vejle, Denmark (Unknown); Hospital of Southern Jutland (Other); Horsens Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAN-FOXY; 2024-517229-18-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-19; First posted 2024-11-29 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2024-11

CONDITIONS: NSTEMI - Non-ST Segment Elevation Myocardial Infarction (MI); Acute Myocardial Infarction (AMI)
Keywords: Acute Myocardial Infarction; Non-ST Segment Elevation Myocardial Infarction; Aspirin; Fondaparinux; Anticoagulation; Coronary Angiography; Percutaneus Coronary Intervention; Acute Coronay Syndrome; Early Invasive Treatment; Refractory ischemia; Bleeding risk; Mortality; Randomized Controlled Trial; New Myocardial Infarction; Non-inferiority Trial; Multicenter Study; Antithrombotic
MeSH Terms: conditions — Ischemia | interventions — Aspirin; Fondaparinux

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, non-inferiority, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin alone (Experimental): Treatment with aspirin alone. The intervention is removal of treatment with fondaparinux
  Interventions: Drug: Aspirin
- Standard Treatment - Aspirin and Fondaparinux (Active Comparator): Standard treatment regime with Aspirin in combination with Fondaparinux.
  Interventions: Drug: Aspirin; Drug: Fondaparinux Sodium

INTERVENTIONS:
Drug: Aspirin — Aspirin bolus of 300 mg followed by 75 mg daily until CAG
Drug: Fondaparinux Sodium — Fondaprinux 2.5 mg subcutaneus daily until CAG (1.5 mg for patients with eGFR 20-50 ml/min/1.73m2)
  Arms: Standard Treatment - Aspirin and Fondaparinux

SUMMARY:
The main goal of this study is to compare two treatments in patients with a specific type of heart attack called Non-ST-elevation Myocardial Infarction (NSTEMI). The investigators want to find out whether using aspirin alone is as effective and safer than using aspirin together with a second blood thinner called fondaparinux.

Both treatments will be given before a scheduled heart procedure called coronary angiography (CAG), which may include balloon dilation and stent placement (PCI) if needed.

The current guidelines recommend using aspirin in combination with a second blood thinner like fondaparinux before CAG and possible PCI. However, these recommendations are based on studies from the 1990s, a time when invasive procedures were not standard practice for these patients. In contrast, nearly all patients with NSTEMI in Denmark (96%) now undergo CAG within 72 hours. This change in practice raises questions about whether the older studies still provide a valid foundation for today's guidelines.

The study aims to answer two questions:

1. Is aspirin alone as effective as aspirin combined with fondaparinux before early CAG and possible PCI?
2. Is aspirin alone safer, with a lower risk of severe bleeding, compared to the combination treatment?

To answer these questions, the investigators will enroll about 5,000 patients with NSTEMI. Participants will be randomly assigned to receive either aspirin alone or aspirin with fondaparinux. The investigators will monitor them for 30 days to compare outcomes such as death, new heart attacks, the need for urgent CAG before the scheduled, and severe bleeding.

DETAILED DESCRIPTION:
Background The current guidelines from European Society of Cardiology (2023) (ESC) and American Heart Association (2014) (AHA) provide a Class-I recommendation for the administration of aspirin together with an anticoagulant in the immediate treatment of Non-ST-Elevation Myocardial Infarction (NSTEMI). For patients scheduled for coronary angiography (CAG) within 24 hours, the recommendation is to initiate unfractionated heparin (UFH) bolus of 70-100 U/kg followed by an adjustable infusion until an activated partial thromboplastin time (APPT) of 60-80 seconds. Patients not planned for CAG within 24 hours are recommended to be treated with fondaparinux 2.5 mg subcutaneous (s.c.) once a day until potential revascularization with percutaneous coronary intervention (PCI) or discharge. According to the clinical guidelines from Danish Society of Cardiology (DSC), fondaparinux is recommended as the first choice for all patients with NSTEMI in Denmark, and heparin is rarely used on this indication.

A plaque rupture in NSTEMI results not only in the activation of platelets but also in the activation of the coagulation cascade through exposure of tissue factor in the extrinsic pathway. This cascade leads to activation of Factor VII and X, which cleave prothrombin to thrombin. Thrombin then converts fibrinogen to fibrin, leading to thrombus formation. Fondaparinux, a synthetic pentasaccharid, directly binds to and enhances the effect of antithrombin, specifically inhibiting activated factor X disrupting the coagulative cascade. Fondaparinux has a half-life of about 17 hours, compared to just 1.5 hours for UFH. This makes the administration and monitoring of UFH treatment substantially more difficult and time-consuming compared to treatment with fondaparinux.

The evidence behind the Class-I recommendation for anticoagulant treatment in patients with NSTEMI is based on two meta-analyses: Oler et al. (1996) and Eikelboom et al. (2000).

The meta-analysis from Oler et al. included six studies that investigated the effect of combination therapy with aspirin and heparin compared with aspirin alone in patients with Non-ST-elevation Acute Coronary Syndrome (NSTEACS), comprising unstable angina pectoris (UAP) and Non-ST-Elevation Myocardial Infarction (NSTEMI). The study showed no statistically significant reduction in the relative risk (RR) = 0.67 (95% CI 0.44-1.02) for new myocardial infarction (MI) or death. However, the results indicated a trend towards a potential positive effect of the combination treatment with both heparin and aspirin.

The indication of a possibly positive effect of combination treatment with both aspirin and anticoagulants was further strengthened with the publication of the FRISC I study (1996), which included 1506 patients with NSTEACS. This was twice as many patients as in all the studies included in the meta-analysis by Oler et al. The patients in the FRISC I study were randomized to treatment with either aspirin and placebo or aspirin and dalteparin (low molecular weight heparin [LMWH]). The primary endpoint was the occurrence of death or new MI within 6 days. The results showed a significant reduction in the primary endpoint, with a odds ratio (OR) of 0.37 (95% CI 0.20-0.68, p = 0.001).

Eikelboom et al. expanded the meta-analysis by Oler et al. to include the FRISC-I study (2000). The expanded meta-analysis demonstrated a statistically significant OR of 0.53 (95% CI 0.38-0.73, p<0.001) in favor of combination therapy compared to aspirin alone when considering death and new MI in patients with NSTEACS.

It's important to note that these studies were conducted at a time when invasive evaluation with CAG was not routinely performed in patients with NSTEACS. For instance, the FRISC-I study showed that the total number of revascularizations after 6 days amounted to 0.8 % and this was due to intractable angina despite relevant medication.

Early invasive evaluation in patients with NSTEMI was only introduced after 1999. A cornerstone of this change was the FRISC-II study (1999), which investigated the effect of an early invasive strategy versus medically treatment in patients with NSTEMI. Of the patients in the invasive arm 96% had a CAG performed within 7 days with an median of 4 days. All patients were treated with either LMWH or UFH prior to the CAG or at least five days in the non-invasive arm. Patients treated invasively compared to noninvasively showed a risk reduction in death or new MI after six months with a risk-ratio of 0.78 (95% CI 0.62-0.98, p=0.031). When considered alone, the occurrence of new MI the risk reduction was also significantly reduced. The difference on mortality alone was not reduced significantly, but there was a trend towards reduction in the invasive arm. Furthermore, the occurrence of symptoms and readmissions were halved. Today, early invasive treatment is recommended in all patients with NSTEMI.

In 2006, the OASIS 5 trial, a randomized controlled trial (RCT) of 20.078 patients, demonstrated that treatment with fondaparinux was non-inferior to treatment with enoxaparin (LMWH) in combinations therapy with aspirin in patients with NSTEACS. The primary endpoint was death, new MI or refractory ischemia within 9 days and the study showed a hazard ration of 1.01 (95% CI 0.90-1.13). Interestingly, treatment with enoxaparin was associated with a higher risk of bleeding, long-time mortality and morbidity. These results have been the foundation for the current guidelines by ESC, which recommend treatment with fondaparinux in patients with NSTEMI when CAG and possibly PCI are not available within 24 hours.

Risk of bleeding:

Intuitively, combination therapy with aspirin together with an anticoagulant will increase the bleeding risk compared with aspirin alone. In the meta-analysis from Eikelboom et al. (2000) they demonstrated an increased OR of 1.88 (CI 95% 0.60-5.87, p= 0.28) for severe bleeding when treated with UFH and aspirin compared to aspirin alone. This result was not significant, however, could imply an increased risk of bleeding with combination therapy.

The meta-analysis from Eikelboom et al. did not report results about minor bleedings. However, by reviewing the papers included in the meta-analysis from Eikelboom et al. one by one, a clear tendency towards an increased risk of minor bleedings can be observed. The occurrence of minor bleedings ranges from 6-14 % in the group with combination therapy compared to 0-3 % in the group with aspirin alone. Even though no statistical analysis was performed, the difference in minor bleeding is undoubtably significant.

Severe bleedings involved events such as intracranial bleeding, requirement of blood transfusion, and bleeding resulting in death. Minor bleedings referred to hematomas and bleeding from insertion site, although the accurate definitions of minor and severe bleedings varied from study to study.

A substantial part of the minor bleeding complications was associated with catheterization. This was also observed in the FRISC-II study, where an increased occurrence of bleeding was observed in the invasive arm compared to the non-invasive arm, despite the shorter treatment period with LMWH in the invasive arm.

Rationale:

All the above-mentioned studies were conducted in a period where early invasive treatment by no means were standard practice in the treatment of patients with NSTEMI. In the FRISC-I study, which must be seen as one of the main pillars in the introduction of anticoagulative treatment in the acute setting of NSTEMI, only 0.8% of all the patients were revascularized after 6 days. This stands in substantial contrast in todays practice, where the year rapport from the Danish Heart Registry from 2022 showed that 96% of patients with either NSTEMI or UAP were invasively assessed and potentially revascularized within 72 hours. This must in any case raise questions about the validity of the studies as a basis for the current guidelines in the treatment of NSTEMI.

A reconsideration of the current treatment strategy is further supported by the potential increased risk of bleeding associated with combination therapy compared to aspirin alone. It is therefore natural to question whether we are currently subjecting patients to unnecessary risk with the current treatment regime.

Additionally, reducing the extent of medical treatment for patients with NSTEMI would lead to decreased cost. Furthermore, you would expect a reduced workload at the cardiology departments, especially them using UFH as their first choice for anticoagulant treatment, as it requires close monitoring of the APPT.

Choice of comparators This study will only compare fondaparinux and aspirin versus aspirin alone as this is the standard practice in Denmark. According to AHA guidelines, options for anticoagulation include Enoxaparin, UFH, fondaparinux or bivalirudin. Similarly, ESC recommends using UFH if CAG is performed within 24 hours, and fondaparinux if the procedure is delayed beyond 24 hours. The evidence from prior studies (Eikelboom et al. and Yusuf et al.) showed that the efficacy of UFH is equivalent to LMWH and that fondaparinux is equivalent to LMWH. Based on this, the investigators believe that the results from this study can be applicable to the other options of anticoagulative options prior to CAG in NSTEMI patients and not exclusively to fondaparinux.

Objectives:

Primary objective:

To compare efficacy in patients treated with aspirin alone compared to combination therapy with fondaparinux and aspirin prior to early invasive strategy in patients with NSTEMI.

Secondary objective:

To evaluate and compare the relative bleeding risk associated with the use of aspirin alone and in combination with fondaparinux prior to an invasive strategy in patients with NSTEMI

Hypothesis's:

* Treatment with aspirin alone is non-inferior in prevention of death, new MI and refractory ischemia within 30 days compared to combination treatment with aspirin and fondaparinux in patients with NSTEMI prior to early invasive strategy
* Treatment with aspirin alone is superior to combination treatment with aspirin and fondaparinux regarding the risk of bleeding defined as BARC above 3 criteria (19)) in patients with NSTEMI prior to early invasive strategy

Sample Size:

According to the annual report from Danish Heart Registry (2022), patient with NSTEACS who underwent PCI had a 30-day mortality rate of 2.1 %. However, this data also includes patients with UAP and patients who was not treated with PCI. The investigators expect the 30-day mortality and 30-day new MI in a cohort with only NSTEMI patients to be slightly higher, around 3 %.

A local review of the data on patients with NSTEMI in Region Midtjylland showed that about 9% these patients were scheduled for an acute CAG after admission. Approximately half of these were assessed as possible subjects to this study.

Based on this, the investigators expect about 5 % of the subjects scheduled for a subacute CAG to convert to acute CAG. In total, this gives us an expected composite event rate of 8%.

The study will require a power of 80% and set a one-sided 97.5 % confidence interval (equivalently to a 95% two-sided confidence interval). Our absolute non-inferiority margin with an expected event rate of 8 % will be 2.2 %. This corresponds to a relative non-inferiority margin of 1.275.

Assuming that the composite event rate is the same in both groups and there truly is no difference between the two interventions, a total of 4776 (2388 in each group) patients are required. This sample size will ensure that the upper limit of a one-sided 97.5%-confidence interval with 80% certainty will exclude a difference of more than 2.2 % in favor of the aspirin group.

Adjustment sample size for loss and interim analysis:

By adjusting for an expected loss of 5 %, our new sample size is 5028. Additionally, to account for one interim analysis, a multiplication factor of 1.008 is applied, resulting in a total sample size of 5068 patients (2534 in each group).

Plans for assessment and collection primary outcome:

The data for assessment of primary endpoints and safety endpoints will mainly be obtained directly from the patient's electronic medical journal. The data will be obtained by study nurses or principal investigators and recorded in a predefined eCRF in REDCap/Corolog. This will include conversion to acute CAG, 30-day mortality, new MI within 30 days, CVA, Severe thrombotic event and severe bleedings as listed under outcomes. These endpoints will be obtained after 30 days. The primary endpoint of 30-day mortality will also be verified through the Danish Civil Registration System to cross-check for any delays or discrepancies in the reporting of deaths in the patients' electronic medical records.

Plans for assessment and collection of secondary outcome, baseline, and other trial data:

Secondary outcomes together with baselines characteristic will be obtained solely from Danish registries.

Location:

All cardiology departments or emergency departments in Denmark with admission of patients with NSTEMI are invited to participate.

Data Safety Monitoring Board (DSMB) - not assigned yet:

The DSMB will be composed of the following members:

* Two cardiologists not involved in the conduct of the trial
* Statistician
* Epidemiologist

The primary role of DSMB is to monitor the safety and efficacy of the trial. The members of DSMB will be independent and will not be involved in the otherwise conduction of the trial or have any financial interests in the outcome of the study. They will be responsible for conduction of the interim analysis.

The DSMB will report directly to the study sponsor, principal investigator and steering committee.

Research ethics and approval:

The trial will be approved through the Clinical Trial Information System (CTIS) by the Medical Ethics Committee (VMK) and the DKMA before initiation.

Publication:

The study expects to result in a publication in at least one recognized international peer-reviewed journal. The paper will be drafted irrespective of whether the results are neutral, positive, negative or inconclusive.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NSTEMI verified by:

  * Rise or/and fall in cardiac troponin (cTN) and
  * Symptoms of acute ischemia or ECG-changes compatible with acute ischemia.
* Age above 18 years old
* Expected remaining lifespan above 1 year
* Informed consent

Exclusion Criteria:

* Treatment with any anticoagulants before enrollment and randomization

  * Including any direct anticoagulant (DOAC), LMWH, UFH or warfarin.
* Not possible with CAG and PCI within 72 hours
* Unsuitable for CAG and possible PCI due to poor condition
* Estimated glomerular filtration rate (eGFR) < 20 ml/min/1.73m2
* Known liver disease
* Active bleeding or high risk of bleeding where treatment with Fondaparinux is contraindicated.
* Anemia (B-Hemoglobin < 6.0 mmol/l)
* Pregnancy or breastfeeding
* Endocarditis
* Indication for acute CAG before enrollment and randomization:

  * ST-elevation Myocardial Infarction (STEMI)
  * Patients classified as "Very High Risk" according to ESC guidelines, defined as(1):

    * Hemodynamic instability (in need of inotropic support) or cardiogenic shock (DANGER-SHOCK criteria (20)) at time of admission.
    * Acute heart failure because of presumed acute ischemia
    * Life-threatening arrhythmias or cardiac arrest
    * Mechanical complications (such as papillary muscle rupture with acute mitral regurgitation, free wall rupture and interventricular rupture)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5076 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of mortality, new myocardial infarction, and clinical deterioration resulting in acute CAG | The primary endpoints will be assessed after day 30.
  Composite of 30-day mortality, 30-day new MI, and clinical deterioration resulting in acute CAG. The endpoints will be assessed through review of the patient's medical journal.
  New Myocardial infarction (MI): Defined as a new MI after the early invasive strategy.
  Clinical deterioration resulting in acute CAG: Defined as conversion to acute coronary angiography (CAG) before the scheduled. Indication for acute CAG is based on the ESC guidelines of "very high risk" NSTEMI (1):

SECONDARY OUTCOMES:
All-cause mortality | Up to 10 years
  Assessed through danish registries
New Myocardial Infarction | Up to 10 years
  Assessed through danish registries
Cerebrovascular accident (CVA) | Up to 30 days
  Including ischemic stroke and Transient Ischemic Attack. Assessed through Danish registries
Length of hospital stay | Up to 30 days
  From admission to discharge at enrollment. Will be assessed through registries and patients medical journal.
Left Ventricular Ejection Fraction at Discharge | Up to 30 days
  Last echocardiography before discharge. From the admission where enrollment took place. Will be assessed from the patients medical journal.

OTHER OUTCOMES:
Severe bleeding | Up to 30 days
  Safety Endpoint:
  Incidence of severe bleeding defined as BARC criteria equal or above 3 within 30 days.
Severe thrombotic event | Up to 30 days
  Safety endpoint:
  Incidence of severe thrombotic events within 30 days including acute MI and CVA

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Department of Cardiology, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
In accordance with Danish and European data protection law

REFERENCES:
- [Background] Kvalitetsudviklingsprogram RK. Dansk Hjerteregister - Årsrapport 2022. 2022.
- [Background] Ashkan E, Pedersen CK, Høfsten DE, et al. Behandlingsvejledning I Akut Koronart Syndrom Dansk Cardiologisk Selskab.
- [Background] Moller JE, Engstrom T, Jensen LO, Eiskjaer H, Mangner N, Polzin A, Schulze PC, Skurk C, Nordbeck P, Clemmensen P, Panoulas V, Zimmer S, Schafer A, Werner N, Frydland M, Holmvang L, Kjaergaard J, Sorensen R, Lonborg J, Lindholm MG, Udesen NLJ, Junker A, Schmidt H, Terkelsen CJ, Christensen S, Christiansen EH, Linke A, Woitek FJ, Westenfeld R, Mobius-Winkler S, Wachtell K, Ravn HB, Lassen JF, Boesgaard S, Gerke O, Hassager C; DanGer Shock Investigators. Microaxial Flow Pump or Standard Care in Infarct-Related Cardiogenic Shock. N Engl J Med. 2024 Apr 18;390(15):1382-1393. doi: 10.1056/NEJMoa2312572. Epub 2024 Apr 7. PMID 38587239
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Cohen M, Adams PC, Parry G, Xiong J, Chamberlain D, Wieczorek I, Fox KA, Chesebro JH, Strain J, Keller C, et al. Combination antithrombotic therapy in unstable rest angina and non-Q-wave infarction in nonprior aspirin users. Primary end points analysis from the ATACS trial. Antithrombotic Therapy in Acute Coronary Syndromes Research Group. Circulation. 1994 Jan;89(1):81-8. doi: 10.1161/01.cir.89.1.81. PMID 8281698
- [Background] Gurfinkel EP, Manos EJ, Mejail RI, Cerda MA, Duronto EA, Garcia CN, Daroca AM, Mautner B. Low molecular weight heparin versus regular heparin or aspirin in the treatment of unstable angina and silent ischemia. J Am Coll Cardiol. 1995 Aug;26(2):313-8. doi: 10.1016/0735-1097(95)80001-w. PMID 7608429
- [Background] Theroux P, Ouimet H, McCans J, Latour JG, Joly P, Levy G, Pelletier E, Juneau M, Stasiak J, deGuise P, et al. Aspirin, heparin, or both to treat acute unstable angina. N Engl J Med. 1988 Oct 27;319(17):1105-11. doi: 10.1056/NEJM198810273191701. PMID 3050522
- [Background] Cohen M, Adams PC, Hawkins L, Bach M, Fuster V. Usefulness of antithrombotic therapy in resting angina pectoris or non-Q-wave myocardial infarction in preventing death and myocardial infarction (a pilot study from the Antithrombotic Therapy in Acute Coronary Syndromes Study Group). Am J Cardiol. 1990 Dec 1;66(19):1287-92. doi: 10.1016/0002-9149(90)91155-y. PMID 2244556
- [Background] Fifth Organization to Assess Strategies in Acute Ischemic Syndromes Investigators; Yusuf S, Mehta SR, Chrolavicius S, Afzal R, Pogue J, Granger CB, Budaj A, Peters RJ, Bassand JP, Wallentin L, Joyner C, Fox KA. Comparison of fondaparinux and enoxaparin in acute coronary syndromes. N Engl J Med. 2006 Apr 6;354(14):1464-76. doi: 10.1056/NEJMoa055443. Epub 2006 Mar 14. PMID 16537663
- [Background] Eikelboom JW, Anand SS, Malmberg K, Weitz JI, Ginsberg JS, Yusuf S. Unfractionated heparin and low-molecular-weight heparin in acute coronary syndrome without ST elevation: a meta-analysis. Lancet. 2000 Jun 3;355(9219):1936-42. doi: 10.1016/S0140-6736(00)02324-2. PMID 10859038
- [Background] Oler A, Whooley MA, Oler J, Grady D. Adding heparin to aspirin reduces the incidence of myocardial infarction and death in patients with unstable angina. A meta-analysis. JAMA. 1996 Sep 11;276(10):811-5. PMID 8769591
- [Background] Cook BW. Anticoagulation management. Semin Intervent Radiol. 2010 Dec;27(4):360-7. doi: 10.1055/s-0030-1267849. PMID 22550377
- [Background] Schiele F. Fondaparinux and acute coronary syndromes: update on the OASIS 5-6 studies. Vasc Health Risk Manag. 2010 Apr 15;6:179-87. doi: 10.2147/vhrm.s6099. PMID 20407625
- [Background] Palta S, Saroa R, Palta A. Overview of the coagulation system. Indian J Anaesth. 2014 Sep;58(5):515-23. doi: 10.4103/0019-5049.144643. PMID 25535411
- [Background] Zaman AG, Helft G, Worthley SG, Badimon JJ. The role of plaque rupture and thrombosis in coronary artery disease. Atherosclerosis. 2000 Apr;149(2):251-66. doi: 10.1016/s0021-9150(99)00479-7. PMID 10729375
- [Background] Bhatt DL, Hulot JS, Moliterno DJ, Harrington RA. Antiplatelet and anticoagulation therapy for acute coronary syndromes. Circ Res. 2014 Jun 6;114(12):1929-43. doi: 10.1161/CIRCRESAHA.114.302737. PMID 24902976
- [Background] Amsterdam EA, Wenger NK, Brindis RG, Casey DE Jr, Ganiats TG, Holmes DR Jr, Jaffe AS, Jneid H, Kelly RF, Kontos MC, Levine GN, Liebson PR, Mukherjee D, Peterson ED, Sabatine MS, Smalling RW, Zieman SJ. 2014 AHA/ACC Guideline for the Management of Patients with Non-ST-Elevation Acute Coronary Syndromes: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2014 Dec 23;64(24):e139-e228. doi: 10.1016/j.jacc.2014.09.017. Epub 2014 Sep 23. No abstract available. PMID 25260718
- [Background] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J. 2023 Oct 12;44(38):3720-3826. doi: 10.1093/eurheartj/ehad191. No abstract available. PMID 37622654
- [Derived] Fur CB, Olsen NT, Lassen JF, Eftekhari A, Stengaard C, Pedersen CK, Rasmussen MB, Terkelsen CJ. Design and rationale of aspirin versus aspirin and fondaparinux prior to early invasive strategy in patients with NSTEMI: The FOXY trial. Am Heart J. 2026 Feb;292:107274. doi: 10.1016/j.ahj.2025.09.006. Epub 2025 Sep 11. PMID 40945808